CLINICAL TRIAL: NCT01639781
Title: Age-dependent Effects of Flavanol Metabolism and Absorption on Vascular Status After Acute and Chronic Application.
Brief Title: Age-dependent Effects of Flavanols on Vascular Status
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: University of Reading (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Klinik für Kardiologie, Pneumologie und Angiologie, Heinrich-Heine University, Duesseldorf
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AGE-111-CH; FLA-111-CH (Other: Flaviola)
Record Dates: First submitted 2012-06-06; First posted 2012-07-13 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Cardiovascular Diseases
Keywords: flavanols; age related cardiovascular effects
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- flavanol rich intervention (Active Comparator): flavanol rich drink
  Interventions: Dietary Supplement: Flavanol rich intervention
- flavanol free intervention (Placebo Comparator): flavanol free drink
  Interventions: Dietary Supplement: Flavanol free control

INTERVENTIONS:
Dietary Supplement: Flavanol rich intervention — Flavanol intervention drinks contain (400 mg flavanols) flavanol rich drink 2 x 400 mg 2 times a day over 2 weeks
  Arms: flavanol rich intervention
Dietary Supplement: Flavanol free control — Calorically, micro- and macronutrient matched control drink free of flavanols flavanol free drink 2 times a day over 2 weeks
  Arms: flavanol free intervention

SUMMARY:
Epidemiological studies suggest that certain foods rich in flavanols, including cocoa products, red wine, and tea, are associated with decreased cardiovascular mortality and morbidity. Dietary interventional studies have corroborated this finding and showed that flavanols can acutely and after sustained ingestion improve surrogate markers of cardiovascular risk including endothelial function. Endothelial dysfunction is the key event in the development and progression of cardiovascular disease. Aging is the major non-modifiable cardiovascular risk factor associated with progressive decline in endothelial function, vascular stiffening and increase in blood pressure. We hypothesize that flavanols can counteract age-dependent vascular changes by interacting with key mechanisms, most prominently endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* healthy male participants between 18-35 years
* healthy male participants between 50-80 years

Exclusion Criteria:

* acute inflammation
* cardiac arrhythmia
* renal failure
* heart failure (NYHA II-IV)
* diabetes mellitus
* CRP > 1 mg/dl
* malignant disease

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Endothelial function | change in flow mediated dilatation between first treatment at day 0 and after last treatment at day 14
  Flow mediated dilatation (FMD)

SECONDARY OUTCOMES:
Plasma flavanol metabolites | analysis of metabolites between first treatment at day 0 and after last treatment at day 14
  Measured by HPLC
Ambulatory blood pressure | blood pressure at day 0 and at day 14
  automatical measurements
Pulse wave velocity | 14 days
  Measured by SphygmoCor
Microvascular function | 14 days
  Measured by Laserdoppler perfusion imaging (LDPI)
Augmentation index | 14 days
  Measured by SphygmoCor
Heart rate | 14 days
  Measured by ECG
Erythrocyte deformability | 14 days
  Measured by Laser-assisted Optical Rotation Cell Analyzer (LORCA)
NO bioavailability | 14 days
  Measured by CLD

CONTACTS AND LOCATIONS:
Overall Officials: Christian Heiss, MD, Principal Investigator — Division of Cardiology, Pulmonology and Vascular Medicine; Malte Kelm, MD, Study Chair — Division of Cardiology, Pulmonology and Vascular Medicine
Locations (1):
- Division of Cardiology, Pulmonology and Vascular Medicine, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Heiss C, Sansone R, Karimi H, Krabbe M, Schuler D, Rodriguez-Mateos A, Kraemer T, Cortese-Krott MM, Kuhnle GG, Spencer JP, Schroeter H, Merx MW, Kelm M; FLAVIOLA Consortium, European Union 7th Framework Program. Impact of cocoa flavanol intake on age-dependent vascular stiffness in healthy men: a randomized, controlled, double-masked trial. Age (Dordr). 2015 Jun;37(3):9794. doi: 10.1007/s11357-015-9794-9. Epub 2015 May 27. PMID 26013912